CLINICAL TRIAL: NCT04360070
Title: The Application of Ketamine for Sedation in Patients With Cardiac Arrest: Feasibility, Safety, and Potential Impact on Neurological Outcomes
Brief Title: The Application of Ketamine for Sedation in Patients With Cardiac Arrest - - KetCat (KETamine in Cardiac ArresT) Study
Acronym: KetCat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, George Medvedev, Head of Neurology, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Ketamine; Neurologic Manifestations
Keywords: Pilot Study; Single-Centre
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Neurologic Manifestations | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Arm (Experimental): Patients randomized to the ketamine arm will receive ketamine as part of their sedation medications during their cardiac arrest treatment
  Interventions: Drug: Ketamine Hydrochloride
- Control Arm (No Intervention): Patients randomized to the control arm will not receive ketamine as part of their sedation medications during their cardiac arrest treatment.

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Parenteral General Anesthetic
  Arms: Ketamine Arm

SUMMARY:
Recent evidence suggests ketamine may attenuate harmful cellular cascades taking place after brain injury that result in permanent damage. The investigators are interested in researching the application of this in the setting of cardiac arrest. Following cardiac arrest, the brain is deprived oxygen for a period of time, leading to the imitation of these harmful cellular processes. The investigators hypothesize that patients who receive ketamine as part of their standard sedation procedures during cardiac arrest treatment have better neurological functioning compared to those who do not.

ELIGIBILITY:
Inclusion Criteria:

* All out-of-hospital cardiac arrests (OHCA) with a "shockable rhythm" (ventricular fibrillation, pulseless ventricular tachycardia) that present to the Royal Columbian Hospital. The patient may be either in active cardiac arrest with shockable rhythm or may have achieved Return of Spontaneous Circulation (ROSC).
* Over 19 years of age
* Patients requiring sedation based on the assessment of the resuscitating physician.

Exclusion Criteria:

* Any other type of cardiac arrest
* Any history of previous, pre-existing neurological deficit
* Started on Extracorporeal Membrane Oxygenation (ECMO)
* Duration of cardiac arrest without ROSC is greater than 30 consecutive minutes
* Known contraindication or hypersensitivity to ketamine
* Awake patient or no standard sedation or no intubation required
* Inability to obtain deferred consent
* Currently enrolled in any other research study involving drugs or devices
* Patients who are pregnant
* Patients who are prisoners
* Patients residing in Long Term Care (LTC) facilities

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12-09 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility Data | through study completion, an average of 6 months.
  To test the appropriateness of the eligibility criteria by recording enrolment rates of eligible patients, test the randomization assignment procedures by evaluating for any difference in baseline characteristics between groups, and test adequate adherence to protocol by recording time taken to administer intervention during sedation procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Fraser Health Authority - Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No